CLINICAL TRIAL: NCT00312429
Title: Cord Blood Transplantation in Adult Recipients
Brief Title: Umbilical Cord Blood Stem Cell Transplantation in Adults With Advanced Blood Disorders or Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2166; R01HL062095-06 (NIH)
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Hematologic Neoplasms
Keywords: Hematological Malignancies; Leukemia; Lymphoma; Myelodysplasia; Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Anemia, Refractory, with Excess of Blasts; Multiple Myeloma | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stem Cell Transplantation — Allogeneic umbilical cord blood stem cell transplant

SUMMARY:
Umbilical cord blood is an important source of stem cells and can be used to treat blood and immune system disorders and certain types of cancer. Stem cell transplants of umbilical cord blood have been shown to be effective in treating illness in children, but more research is needed to confirm the benefit of this procedure in adults. The purpose of this study is to examine the immune system response to cord blood stem cell transplantation in adults with advanced blood disorders or cancer.

DETAILED DESCRIPTION:
The use of umbilical cord blood stem cells to treat blood disorders and cancer is an important medical advance; currently, more than 45 disorders can be treated with this method. While bone marrow transplants are the most common method for stem cell donations, research has shown that there are many advantages to using allogeneic grafts of stem cells obtained from umbilical cord blood. Cord blood stem cells are relatively easy to obtain. Additionally, a perfect donor match is not necessary, thereby decreasing the likelihood of graft-versus-host disease (GVHD), a serious side effect in which donor stem cells attack the recipient's tissues. Cord blood has been used successfully in pediatric patients but its benefit in adults remains untested. The purpose of this study is to evaluate the effectiveness of umbilical cord blood stem cell transplantation in adults with advanced blood disorders or cancer. Upon receiving an allogeneic stem cell transplant using umbilical cord blood, participants will be observed for successful engraftment in which the transplanted stem cells "take" and begin producing new blood cells. The incidence of GVHD and the overall immune system's response will also be examined. In turn, these findings may guide future umbilical cord blood stem cell clinical trials.

This 1-year study will enroll individuals with advanced blood diseases or cancer. Participants will receive an allogeneic umbilical cord blood stem cell transplant and will be closely monitored while in the hospital to determine when engraftment occurs and if GVHD develops. Study visits will occur at Months 1, 2, 3, 6, 9, and Year 1. At each visit, participants will have blood drawn for laboratory testing and for evaluation of immune system response. Quality of life questionnaires will also be completed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis reviewed at transplant center and confirmed to fit the criterion for high risk blood disease or cancer, as defined for the study
* Estimated life expectancy of at least 6 weeks following study entry
* Cancer and Leukemia Group B (CALGB) performance status less than or equal to 2
* White blood cell count, platelet, hematocrit, tuberculosis, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, creatinine, and HIV test results reviewed by transplant center
* Multiple gated acquisition (MUGA), echocardiogram, cardiac MRI, and/or pulmonary function tests (PFT) performed and reviewed by transplant center (for individuals with an ejection fraction and diffusing capacity [DLCO] of 40-50%, the appropriate cardiology or pulmonary consultations should be considered if the individual has severe heart or lung disease at the initiation of therapy)
* Sufficient number of umbilical cord blood units available for transplantation
* If female, willing to use contraception throughout the study

Exclusion Criteria:

* Undergoing Interleukin-2 (IL-2) therapy within 8 weeks of study entry
* Diagnosed with a medical or psychiatric illness that may interfere with study participation
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2002-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

SECONDARY OUTCOMES:
Survival Rates | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Nelson J. Chao, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States